CLINICAL TRIAL: NCT05368194
Title: The FEASST Study: Food Intake and Epigenetic Alteration in the Spermatozoa of Singletons and Twins
Brief Title: Food Intake and Epigenetic Alteration in the Spermatozoa of Singletons and Twins
Acronym: FEASST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Deakin University (Other); Monash Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-20061598
Record Dates: First submitted 2021-12-16; First posted 2022-05-10 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Fertility Issues; Nutrition, Healthy; Epigenetic Disorder; Overnutrition
MeSH Terms: conditions — Infertility; Overnutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isocaloric Arm (Experimental): Participants within the isocaloric arm will be provided with food provisions in accordance with their nutrition needs. Participants within this arm will be further randomised to the order of first and second dietary interventions for the crossover design; unprocessed diet or processed diet.
  Interventions: Dietary Supplement: Isocaloric Unprocessed Diet; Dietary Supplement: Isocaloric Processed Diet
- Excess Calorie Arm (Experimental): Participants within the excess calorie arm will be provided with food provisions in accordance with their nutrition needs plus an additional 500 kilocalories per day. Participants within this arm will be further randomised to the order of first and second dietary interventions for the crossover design; unprocessed diet or processed diet.
  Interventions: Dietary Supplement: Excess Calorie Unprocessed Diet; Dietary Supplement: Excess Calorie Processed Diet

INTERVENTIONS:
Dietary Supplement: Isocaloric Unprocessed Diet — Intervention consists of an unprocessed diet meeting the Nordic and Australian Dietary Guidelines for food groups and micronutrients, wherein participants will be supplied with food providing kilocalories (kcal) in accordance with their nutritional needs as calculated based on theSchofield equation based on their weight, activity multiplier, and age at baseline. Almost all food and beverage products provided during this treatment to fall into the category of unprocessed/minimally processed foods and processed culinary ingredients in accordance with the NOVA classification system.
  Arms: Isocaloric Arm
Dietary Supplement: Isocaloric Processed Diet — Intervention consists of a processed diet based on the dietary intake pattern resembling a processed western dietary intake pattern representative of the typical intake pattern of American men aged 19- 50, wherein participants will be supplied with food providing kcals in accordance with their nutritional needs as calculated based on the Schofield equation based on their height, weight, activity multiplier, and age at baseline. Almost all food and beverage products provided during this treatment to fall into the category of processed foods and ultra-processed foods in accordance with the NOVA classification system.
  Arms: Isocaloric Arm
Dietary Supplement: Excess Calorie Unprocessed Diet — Intervention consists of an unprocessed diet meeting the Nordic and Australian Dietary Guidelines for food groups and micronutrients, wherein participants will be supplied with food providing kilocalories (kcal) in accordance with their nutritional needs as calculated based on theSchofield equation based on their weight, activity multiplier, and age at baseline, plus an excess of 500 kcal per day. Almost all food and beverage products provided during this treatment to fall into the category of unprocessed/minimally processed foods and processed culinary ingredients in accordance with the NOVA classification system.
  Arms: Excess Calorie Arm
Dietary Supplement: Excess Calorie Processed Diet — Intervention consists of a processed diet based on the dietary intake pattern resembling a processed western dietary intake pattern representative of the typical intake pattern of American men aged 19- 50, wherein participants will be supplied with food providing kcals in accordance with their nutritional needs as calculated based on the Schofield equation based on their height, weight, activity multiplier, and age at baseline, plus an excess of 500 kcal per day. Almost all food and beverage products provided during this treatment to fall into the category of processed foods and ultra-processed foods in accordance with the NOVA classification system.
  Arms: Excess Calorie Arm

SUMMARY:
The purpose of this study is to elucidate the role of acute dietary intake in male populations, and its impact on spermatozoa quality, integrity, content and epigenetic programming.

DETAILED DESCRIPTION:
The FEASST study has been designed to determine the impact of diet on the content, quality, and genetic programming of sperm. They are specifically interested in determining if a man's diet plays a role in influencing the health of his potential, future offspring through modifications of the sperm. Previous research has highlighted that certain dietary patterns in fathers-to-be may lead to variable health outcome for their children. However, the specific effect of a man's diet has yet to be fully understood. This study will help understand the impact of a man's diet on semen quality and potential downstream implications for child health, to aid in the development of dietary guidelines for future fathers-to-be.

For this study, male participants will be provided with two prescribed diets for three-week increments punctuated by a three month break. Health information and biological samples such as blood, semen, and saliva will be collected from study participants throughout the five month period. The diets will consist of a 'Processed diet', mimicking a traditional Western dietary intake pattern and an 'Unprocessed diet', based upon current dietary guidelines at quantities either adequate for the participants energetic needs or 500 calories in excess per day.

Patient information and samples will be collected before and after each dietary intervention. Aspects of patient health examined at various time points include weight, body fat percentage, sperm quality, epigenetic sequencing, serum levels of metabolic parameters, and survey information surrounding health history, typical diet, physical activity patterns, and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 20 to 35 years old
* BMI 18.5 to 30
* Located within the Copenhagen region
* Fluent in English and/or Danish language
* Sperm concentration of >15 mil/mL according to the WHO's criteria for semen quality
* Semen volume of >1.5mL mL according to the WHO's criteria for semen quality
* Clinician approval for participation in study
* Obtained informed consent

Exclusion Criteria:

* Self-reported history of serious or chronic illness
* Self-reported history of Obesity
* History of any food restrictions
* History of allergies to any food products
* History of disordered eating
* Record of current use of drugs, alcohol (>14 units per week and/or chronic binge drinking), and/or tobacco/nicotine products within the past month
* Current use of prescription medication
* Engage in > 200 minutes of vigorous aerobic exercise per week
* Currently actively trying to conceive a child
* Diagnosis of infertility or disease of the reproductive system
* Evidence of dysregulated metabolism, characterized by the occurrence of any one of the following:

  * Waist circumference >102 cm
  * Blood pressure > 130/85 mm Hg

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Spermatozoa DNA Methylation via Reduced Representation Bisulfite Sequencing | 3 weeks
  Differential methylation of CpG sites within mature spermatozoa determined from extracted genomic DNA which has undergone library preperation with Ovation® RRBS Methyl-Seq (NuGEN Technologies) and sequenced on a NextSeq Illumina platform.

SECONDARY OUTCOMES:
Sperm Concentration | 3 weeks
  Measured in million sperm per mL using LensHooke X1 Pro Semen Quality Analyser and Microscopy-based methodology
Semen Volume | 3 weeks
  Measured in mL assuming the density of semen to be 1 g/ml
Sperm Motility | 3 weeks
  Measured in precent of sperm classified as progressively motile and non-progressively motile using LensHooke X1 Pro Semen Quality Analyser and Microscopy-based methodology
Spermatozoa smallRNA expression via sequencing of total smallRNA species | 3 weeks
  Differential expression of small RNA species within mature spermatozoa performed by generation of RNA sequencing libraries using NEXTFLEX® Small RNA-Seq Kit for Illumina (PerkinElmer), according to the manufacturer's instructions, and sequenced on a NextSeq Illumina platform.
Weight | 3 weeks
  Measured in kilograms using a scale (Tanita DC 430 SMA)
Body Mass Index (BMI) | 3 weeks
  Calculated based on height and weight measurement using the equation BMI=kg/m^2
Waist Circumference | 3 weeks
  Measured in centimetres using a flexible measuring tape (SECA Measuring Tape 201 cm)
Hip Circumference | 3 weeks
  Measured in centimetres using a flexible measuring tape (SECA Measuring Tape 201 cm)
Body Fat Precentage | 3 weeks
  Measured using DEXA Scanner and Software (GE Lunar Prodigy)
C-reactive protein (CRP) | 3 weeks
  Measured in milligrams per litre in serum
Lipoproteins | 3 weeks
  Measuring high density lipoproteins and low density lipoproteins in milligrams per litre in plasma
Total protein | 3 weeks
  Measured in grams per litre in serum
Testosterone | 3 weeks
  Measured in nanograms per deciliter in plasma
Follicle stimulating hormone (FSH) | 3 weeks
  Measured in international units per milliliter in serum
Luteinizing hormone (LH) | 3 weeks
  Measured in international units per liters in plasma
Progesterone | 3 weeks
  Measured in nanograms per milliliter in serum
Estradiol | 3 weeks
  Measured in picograms per milliliter in serum
Oestradiol | 3 weeks
  Measured in picograms per milliliter in serum
Fasting Blood Glucose | 3 weeks
  Measured in whole blood using a handheld glucometer and test strip (Contour next Blood Glucose Meter and Blood Sugar Test strip)
Insulin | 3 weeks
  Measured in microunits per milliliter in serum
Haemoglobin A1c (HbA1c) | 3 weeks
  Measured in mmol/mol in plasma
Blood pressure | 3 weeks
  Systolic and Diastolic blood pressure measured in mmHg using an automatic blood pressure cuff (Omron M6 Comfort Automatic Upper Arm Blood Pressure Monitor, 22-42cm)
Leptin | 3 weeks
  Measured in ng/mL in plasma
Glucagon-like peptide 1 (GLP-1) | 3 weeks
  Measured in pmol/L in plasma
Gastric inhibitory peptide (GIP) | 3 weeks
  Measured in pg/mL in serum
Glucagon | 3 weeks
  Measured in pg/mL in serum
Ghrelin | 3 weeks
  Measured in pg/mL in plasma
Fibroblast growth factor 21 (FGF-21) | 3 weeks
  Measured in pg/ml in serum
Peripheral blood mononuclear cell (PBMC) DNA methylation via Reduced Representation Bisulfite Sequencing | 3 weeks
  Differential methylation of CpG sites within PBMCs determined from extracted genomic DNA which has undergone library preperation with Ovation® RRBS Methyl-Seq (NuGEN Technologies) and sequenced on a NextSeq Illumina platform.

CONTACTS AND LOCATIONS:
Overall Officials: Romain Barrès, PhD, Principal Investigator — University of Copenhagen Novo Nordisk Foundation Center for Basic Metabolic Research
Locations (1):
- University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No